CLINICAL TRIAL: NCT06819891
Title: A Phase III, Multicenter, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Induction Therapy With RO7790121 in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Assess the Efficacy and Safety of Induction Therapy With Afimkibart (RO7790121) in Participants With Moderately to Severely Active Crohn's Disease
Acronym: SIBERITE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA45332; 2024-513054-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Moderately to Severely Active Crohns Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afimkibart (Experimental): Participants will receive afimkibart intravenously (IV) followed by afimkibart subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Placebo (Placebo Comparator): Participants will receive placebo IV followed by afimkibart SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as IV infusion. Afimkibart will be administered as SC injection.
  Other Names: PF-06480605; RVT-3101; RG6631; RO7790121
  Arms: Afimkibart
Drug: Placebo — Placebo matching IV afimkibart.
  Arms: Placebo

SUMMARY:
This Phase III, multicenter, double-blind, placebo-controlled study will evaluate the efficacy and safety of induction therapy with Afimkibart (also known as RO7790121) in participants with moderately to severely active Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD
* Moderately to severely active CD
* Bodyweight >= 40 kilogram (kg)
* Demonstrated inadequate response, loss of response and/or intolerance to at least one protocol-specified conventional or advanced CD therapy
* Males and females of childbearing potential must meet protocol criteria for contraception requirements

Exclusion Criteria:

* Current diagnosis of ulcerative colitis (UC) or indeterminate colitis, ischemic colitis, infectious colitis, radiation colitis, microscopic colitis
* Participant with a history of >= 3 bowel resections (> 2 missing segments of the 5 following segments: terminal ilelium, right colon, transverse colon, sigmoid and left colon, and rectum)
* Diagnosis of short gut or short bowel syndrome
* Presence of an ileostomy, colostomy or ileoanal pouch
* Participants with symptomatic bowel strictures, fulminant colitis, or toxic megacolon
* Presence of abdominal or perianal abscess
* Presence of rectovaginal, enterovaginal, high output enterocutaneous fistula, enterovesical fistulas or perianal fistulas with >3 openings
* Participants with symptomatic bowel strictures, fulminant colitis, or toxic megacolon
* Current diagnosis or suspicion of primary sclerosing cholangitis
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Any past or current evidence of cancer of gastrointestinal tract, definite low-grade or high-grade colonic dysplasia
* History of non-gastrointestinal cancer, with the exception of adequately treated non-metastatic basal cell or squamous cell skin cancer or in situ cervical cancer
* Evidence of infection with Clostridioides difficile (C. difficile; formerly known as Clostridium difficile), cytomegalovirus (CMV), human immunodeficiency virus (HIV), Hepatitis B (HBV), Hepatitis C (HCV) during screening
* Has evidence of active tuberculosis (TB), latent TB not successfully treated (per local guidance) or inadequately treated TB
* Has received protocol-specified prohibited medicines, including known exposure to any type of anti-TL1A therapy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission per Crohn's Disease Activity Index (CDAI) Score | At Week 12
  Percentage of participants achieving a CDAI score of <150. The index is a weighted sum of scores on eight components: number of liquid or soft stools (stool frequency), abdominal pain, general well-being, number of complications, use of anti-diarrheal medication, presence of an abdominal mass, hematocrit, and percentage deviation from standard body weight. CDAI generally ranges from 0 to roughly 600, with higher values indicating greater activity.
Percentage of Participants with Endoscopic Response | At Week 12
  Percentage of participants achieving a decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) of >=50% from baseline. The SES-CD is a composite of four features of endoscopic activity (presence and size of ulcers, extent of ulcerated surface, extent of affected and presence and type of narrowings or stenosis) in up to five ileocolonic segments (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum). Each feature is scored on a scale from 0 to 3, giving segment subscores of 0 to 12 points and a total SES-CD range of 0-60, with a higher value indicating greater severity.

SECONDARY OUTCOMES:
Percentage of Participants with Symptomatic Remission | At Week 12
  Percentage of participants with the daily number of liquid or very soft stools <=2.8 and the average of daily abdominal pain scores in the past week <=1, with neither being greater than baseline.
Percentage of Participants with Endoscopic Remission | At Week 12
  Percentage of participants with an SES-CD of 0 to 4 with a decrease from baseline >=2 and no subscore >1.
Percentage of Participants with Ulcer-free Endoscopy | At Week 12
  Percentage of participants with an SES-CD ulcerated surface subscore of 0.
Average of Daily Number of Liquid or Very Soft Stools in the Past Week (SF) | Baseline through Week 12
  Daily average number of liquid or very soft stools over 7 days.
Average of Daily Abdominal Pain Scores in the Past Week (APS) | Baseline through Week 12
  The average daily rating of abdominal pain in the past 7 days. The pain is assessed on a scale of 0-3 with 0 indicating no pain and 3 indicating severe pain.
Bowel Urgency | Baseline to Week 12
  Bowel urgency from baseline through week 12 and. Bowel urgency is a single-item self-reported assessment of sudden or immediate need to have a bowel movement in the past 24 hours. The item response is reported on a 4-point Likert scale, from "None" to "Severe."
Fatigue | Baseline to Week 12
  Fatigue, as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F), from baseline to Week 12. FACIT-F is a 13-item self-reported assessment of fatigue. Each item response option indicates the degree to which a given statement describing the level or impact of fatigue applies in the past 7 days. Response options are graded on a 5-point Likert-type scale, from "Not at all" to "Very much."
Inflammatory Bowel Disease Questionnaire (IBDQ) Score | Baseline to Week 12
  Change in IBDQ score from baseline to week 12. The IBDQ is a 32-item questionnaire that measures four domains: bowel symptoms (10 questions); systemic symptoms (5 questions); emotional function (12 questions); and social function (5 questions). The total score ranges from 32-224, with a higher score indicating a better quality of life.
Percentage of Participants with Clinical Remission: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving a CDAI score of <150 at Week 12 in biomarker-defined subgroups. The index is a weighted sum of scores on eight components: number of liquid or soft stools (stool frequency), abdominal pain, general well-being, number of complications, use of anti-diarrheal medication, presence of an abdominal mass, hematocrit, and percentage deviation from standard body weight. CDAI generally ranges from 0 to roughly 600, with higher values indicating greater activity.
Percentage of Participants with Endoscopic Response: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving a decrease in SES-CD of >=50% from baseline. The SES-CD is a composite of four features of endoscopic activity (presence and size of ulcers, extent of ulcerated surface, extent of affected and presence and type of narrowings or stenosis) in up to five ileocolonic segments (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum). Each feature is scored on a scale from 0 to 3, giving segment subscores of 0 to 12 points and a total SES-CD range of 0-60, with a higher value indicating greater severity.
Percentage of Participants with Clinical Response | At Week 12
  Percentage of participants with a decrease >=100 in CDAI from baseline.
Percentage of Participants with Symptomatic Response | At Week 12
  Percentage of participants with a decrease >=30% in both SF and APS, with neither being greater than baseline.
Overall Change in CD Symptoms | Baseline to Weeks 2, 6 and 12
  Overall change in CD symptoms, as measured by the Patient Global Impression of Change (PGIC) from baseline to Weeks 2, 6 and 12. PGIC measures overall change in Crohn's disease symptoms from "Much better" to "Much worse".
Overall Severity in CD Symptoms | Baseline to Weeks 2, 6 and 12
  Overall severity in CD symptoms, as measured by the Patient Global Impression of Severity (PGIS) from baseline to Weeks 2, 6 and 12. PGIS measures severity of Crohn's disease symptoms from "None" to "Very severe".
Change in General Well-being | Baseline through Week 12
  The average daily rating of general well-being in the past 7 days. Well-being is assessed on a scale of 0-4 with 0 indicating generally well and 4 indicating terrible.
Incidence and Severity of Adverse Events (AEs) | Up to 30 Weeks after Baseline
  Incidence and severity of AEs, including serious AEs, AEs leading to treatment discontinuation and AEs of special interest.
Presence of Draining Fistulas | Baseline through Week 12
  Fistulas will be assessed for draining or closed status, where closed fistulas will be assessed by the investigator as no longer draining.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (149):
- United States (38):
  - Sun City Clinical Research, Glendale, Arizona
  - Om Research LLC, Lancaster, California
  - Hoag Memorial Hospital Presbyterian;Hoag Center for Research and Education, Newport Beach, California
  - Amicis Research Center, Santa Clarita, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - J&A Clinical Research, Doral, Florida
  - Homestead Associates in Research, Inc., Miami, Florida
  - Allied Biomedical Research Institute, Inc, Miami, Florida
  - Rejuvaline Medical Research, Miami, Florida
  - Miami Beach Clinical Research Center, Miami Beach, Florida
  - Eminat Research Group, Miramar, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Louisiana Research Center - GastroIntestinal Associates, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - University of Massachusetts Memorial Medical Center, North Worcester, Massachusetts
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Gastrointestinal Associates Research, Flowood, Mississippi
  - Virtua Crohns and Colitis Center, Moorestown, New Jersey
  - Ellipsis Research Group, Brooklyn, New York
  - Intercity Gastroenterology, Fresh Meadows, New York
  - James J Peters Veterans Affairs Medical Center, The Bronx, New York
  - Digestive Disease Medicine of Central New York, Utica, New York
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Clinical Inquest Center, Beavercreek, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center - Multidisciplinary Spine Clinic - James W. Aston Ambulatory Care Center, Dallas, Texas
  - GI Alliance, Garland, Texas
  - Integrity Advanced Therapeutics PLLC, Houston, Texas
  - Carta - Clinical Associates In Research Therapeutics Of America;LLC, San Antonio, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - University Physicians and Surgeons Inc, dba Marshall Health, Huntington, West Virginia
- Argentina (2):
  - Instituto Medico CER, Quilmes
  - CICE 9 de Julio, San Miguel de Tucumán
- Australia (4):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Coral Sea Clinical Research Institute, Mackay, Queensland
  - Footscray Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (3):
  - CHU St Pierre (St Pierre), Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
- Brazil (6):
  - Instituto Lobus Unimed Volta Redonda, Volta Redonda, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Newdata Clinical Trials, Aracaju, Sergipe
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
- MC " Sveti Ivan Rilski Chudotvorets- 2010, Plovdiv, Bulgaria
- Canada (5):
  - Barrie GI Associates, Barrie, Ontario
  - GNRR Digestive Clinics and Research Center Inc., Brampton, Ontario
  - London Health Sciences Centre Uni Campus, London, Ontario
  - Toronto Immune and Digestive Health Institute, North YORK, Ontario
  - CIUSSS de l Est de l Ile de Montreal - Hopital Maisonneuve Rosemont, Montreal, Quebec
- Centro de Investigación Clínica UC-CICUC, Santiago, Chile
- China (18):
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affilliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Jinhua municipal central hospital, Jinhua, Zhejiang
  - Beijing Union Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - Guangzhou First People's Hospital, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Hainan General Hospital, Haikou
  - Huizhou First Hospital, Huizhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Hebei Medical University - The Second Hospital, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá
  - Clínica de la Mujer, Bogotá
  - Oncomedica S.A., Montería
- Borzan Polyclinic, Osijek, Croatia
- Czechia (5):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Institutu Klinicke a Experimentaini Mediciny (IKEM);Klinika hepatogastroenterologie, Prague
  - ISCARE a.s., Prague
  - Krajska zdravotni, a.s. ? Masarykova nemocnice v Usti nad Labem, o.z., Ocni oddeleni, Ústí nad Labem
- France (11):
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CH Dptal Les Oudairies, La Roche-sur-Yon
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hopital Dupuytren, Limoges
  - Hopital Saint-Eloi, Montpellier
  - Institut des MICI, Clinique Ambroise Paré, Neuilly-sur-Seine
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- Hungary (3):
  - Észak-Pesti Centrumkórház-Honvédkórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Vas-Oxy Egeszsegugyi Kft, Szombathely
- India (7):
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Surat Institute of Digestive Sciences Hospitals, Surat, Gujarat
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - MIDAS Multispeciality Hospital, Nagpur (urban), Maharashtra
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - AIG Hospitals, Gachibowli, Telangana
  - Yashoda Hospitals, Secunderabad, Telangana
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (8):
  - Ospedale Madonna delle Grazie, Matera, Basilicate
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi-Via Massarenti, Bologna, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico Di Roma, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Lombardy
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
- Poland (16):
  - Gastromed Kralisz, Romatowski, Stachurska sp.j., Bia?ystok
  - Medical Center Kermed, Bydgoszcz
  - Szpital Miejski sw. Jana Paw?a II w Elblagu, Elblag
  - Osrodek Badan Klinicznych Bd Research, I?awa
  - MZ Badania Slowik Zymla Sp.j., Knurów
  - Centrum Medyczne Promed, Krakow
  - Medrise sp z o.o, Lublin
  - Clinical Research Center Sp. z o.o. MEDIC-R Spó?ka Komandytowa, Poznan
  - EMC Instytut Medyczny SA, Późna
  - Gabinety Lekarskie Rivermed, Późna
  - Endoskopia Sp. z o.o., Sopot
  - Sonomed Sp. z o.o., Szczecin
  - Centrum Zdrowia-MDM, Warsaw
  - Medon Clinical Research sp. z o.o, Warsaw
  - Vivamed Spolka Z Ograniczona Odpowiedzialnoscia, Warsaw
  - PlanetMed sp. z o.o., Wroc?aw
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital de Santa Maria, Lisbon
  - Hospital de Sao Joao, Porto
  - Centro Hospitalar de Entre Douro e Vouga - H. São Sebastião, Santa Maria da Feira
  - Hospital Sao Teotonio, Viseu
- Slovakia (2):
  - ABAWI spol. s r.o., Bratislava
  - KM Management spol. s r.o., Nitra
- Spain (3):
  - Fundacion Hospital de Alcorcon, Alcorcón, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico Univ. Lozano Blesa, Zaragoza
- United Kingdom (3):
  - Fairfield General Hospital, Bury
  - Bronglais General Hospital, Llanrhystud
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing